CLINICAL TRIAL: NCT02272491
Title: Monolithic Zirconia Crowns for Single Implants in the Molar Region: a Randomized Controlled Clinical Trial
Brief Title: Monolithic Zirconia Crowns for Single Implants in the Molar Region: a Multicenter Clinical Trial
Acronym: MonoZrO2crown
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ITI Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0191
Record Dates: First submitted 2014-10-10; First posted 2014-10-23 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Implant-supported Single Crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZrO2 (Experimental): 1. Straumann CARES Variobase Abutment RN
  2. Straumann CARES Full Contour Zerion HT The monolithic zircona crown (2) will be bonded to the titanium base (1)
  Interventions: Device: ZrO2 (Straumann CARES)
- PFM crown (Active Comparator): Straumann Gold Abutment RN Porcelain-fused-to-metal crown consisting of a gold abutment, a gold core, and veneering ceramic
  Interventions: Device: PFM crown (Straumann Gold)

INTERVENTIONS:
Device: ZrO2 (Straumann CARES) — 1. Straumann CARES Variobase Abutment RN
  2. Straumann CARES Full Contour Zerion HT The monolithic zircona crown (2) will be bonded to the titanium base (1)
  Arms: ZrO2
Device: PFM crown (Straumann Gold) — Porcelain-fused-to-metal crown consisting of a gold abutment, a gold core, and veneering ceramic
  Arms: PFM crown

SUMMARY:
The aim of the present study is to test whether or not the use of translucent monolithic zirconia crowns bonded to a titanium base abutment perform similar to porcelain-fused-to-metal crowns on single implants in the posterior region.

DETAILED DESCRIPTION:
In the majority of studies on implant-supported restorations, a considerable rate of fractures of the veneering ceramic was reported. The clinical data is restricted to full-ceramic implant-supported reconstructions in the anterior region. No clinical data is available on the performance of full-ceramic restorations in the molar region.

The use of translucent monolithic zirconia for implant-supported crowns (without veneering ceramic) may reduce the technical complication rate and allow for sufficient aesthetic results in the molar region. To date, no clinical trial investigating monolithic zirconia crowns for single molar implants is available.

The primary outcome of the study is the technical complication rate. This outcome represents an indicator for the prosthetic success of the implant-supported crown. The main biological secondary outcomes are marginal bone level, histological signs of inflammation, and presence of pathogenic bacteria. Further outcomes are crown survival, wear of the crown and of the antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male and female patients from 18-80 years of age
* Presence of a Straumann Tissue Level implant with a regular platform (4.8 mm diameter platform) in the maxillary or mandibular molar region
* Need for a single implant-supported crown
* Implant position enabling screw-retained crown
* Presence of antagonist

Exclusion Criteria:

* Women who are pregnant at the date of inclusion
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Smoking more than 15 cigarettes a day
* Poor oral hygiene (Plaque Index over 30%)
* Bruxism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Technical complication rate | 5 years
  assessed by USPHS-criteria

SECONDARY OUTCOMES:
Survival rate | 6-month, 1, 3, 5, 7, 10 years
Biological complication rate | 6-month, 1, 3, 5, 7, 10 years
  assessed by bleeding on probing, pocket probing depth, marginal bone level
Wear rate of the antagonist | 6-month, 1, 3, 5, 7, 10 years
  assessed by a volumetric analysis software
Technical complication rate | 6-month, 1, 3 , 7, 10 years
  assessed by USPHS-criteria

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ioannidis, Dr., Principal Investigator — Clinic of Reconstructive Dentistry
Locations (1):
- Clinic of Reconstructive Dentistry, Zurich, Switzerland